CLINICAL TRIAL: NCT06891014
Title: Effects of Regular Exercise on Sensory-motor Functions and Fall Risk in the Elderly
Acronym: FallRisk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus International University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Sıddıka Fatma Uygur, Prof. Dr., Cyprus International University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: -020-1285
Record Dates: First submitted 2025-03-11; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Fall Risk; Exercise; Functional Outcomes; Aging
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Cross-Sectional Case Control
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and assessor will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combine Exercise Group (Active Comparator): Participants who will participate in a combine exercise program under the control of a physiotherapist, 2-3 days a week for 8 weeks.
  Interventions: Other: Combine Exercise
- Control Group (No Intervention): Control Group with a sedentary lifestyle

INTERVENTIONS:
Other: Combine Exercise — The participants in the exercise group will be individuals over the age of 65 who applied the same exercise programs 2-3 days a week for 8 weeks under the control of two different physiotherapists independent of the study. The exercise session will be applied for one hour, including a warm-up phase, a combined exercise program including strengthening, stretching, balance and proprioceptive exercises, and a cool-down phase.
  Other Names: Exercise
  Arms: Combine Exercise Group

SUMMARY:
Falls in elderly population are an important public health problem. The aim of this study is to examine the vibration, proprioception, muscle strength, static balance, reaction time and postural stability parameters of female individuals aged 65 and over who exercise regularly by comparing them with sedentary female individuals in the same age group and to determine the effect rates of these parameters on fall risk. A total of 92 individuals will evaluate in the study, including 46 participants who perform regular exercise and 46 participants with a sedentary lifestyle. Participants who performs regular exercise will determine among individuals who going to participate in a combined exercise program under the control of a physiotherapist, 2-3 days a week for 8 weeks. The socio-demographic characteristics, health conditions and exercise habits of the participants will be recorded. For evaluating the physical activity levels of the participants, the International Physical Activity Questionnaire-short form (IPAQ-SF); for vibration sense evaluation, 128-Hz frequency tuning fork; for the evaluation of proprioception sense, angle repetition test; for the isometric muscle strength assessment, digital hand dynamometer; for static balance evaluation, standing stork balance test; for reaction time evaluation, MoART measuring device; for postural stability evaluation, PROKIN-PK200W* (Tecnobody, Italy) device and for fall risk assessment, Morse fall scale and MAHC-10 fall questionnaire will be used.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary individuals with an International Physical Activity Questionnaire (IPAQ) score of <600 (for control group)
* Individuals who will be participated in an eight-week regular exercise program (for the exercise group)
* Those who scored 24 or higher on the standardized Mini-Mental State Examination, individuals without communication problems, and those who were not bedridden or wheelchair-bound.

Exclusion Criteria:

* Individuals who had received any diagnosis/treatment for spinal or lower extremity problems or had undergone surgery within the last six months, as well as those with severe chronic illnesses or uncontrolled conditions (e.g., hypertension, cancer), will be excluded from the study.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 92 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Fall Risk | Through study completion, an average of 5 months
  Morse Fall Scale (MFS) will be used to assess fall risk. For MFS; A total score between 0-24 indicates a low risk of falling; 25-50 indicates moderate risk of falling, and total score of 51 and above indicates a high risk of falling.
Fall Risk | Through study completion, an average of 5 months
  Missouri Alliance for Home Care (MAHC-10) Fall Risk Assessment Questionnaire will be used to assess fall risk. The MAHC-10 fall risk assessment questionnaire with 10 questions is method for determining the risk of falling in the home environment. The minimum score "0", indicates no risk factors while maximum score "10" indicates that all risk factors are present. A score below 4 indicates no risk of falling, a scores 4 or above indicate high risk of falling.
Vibration Sense | Through study completion, an average of 5 months
  Vibration sense will be assesed from the 1st metatarsal head of the dominant and non-dominant feet using a tuning fork (128 Hz, Mesitas Istanbul, Turkiye). Participants will be asked to start the digital stopwatch in their hand when they felt the vibration and to stop the stopwatch when the vibration ended. The assessment will be repeated three times and the average value will calculate. The values obtained will record in seconds (s). The sensation of vibration felt for more than 10 seconds will be categorized as "normal," felt for 1-9 seconds as "reduced," and felt for less than 1 second as "absent"
Proprioception Sense | Through study completion, an average of 5 months
  Ankle proprioception sense will be evaluated using the angle repetition test. A 180-degree platform drawn at 1° intervals will be used for ankle dorsiflexion and plantar flexion movements. The target angles for the test will be determined as 10° for dorsiflexion movement and 20° for plantar flexion. Before the evaluation, the participants will be asked to perceive that position by passively bringing their feet to the target angles (dorsiflexion: 10°, plantar flexion: 20°). Then, the participants will be asked to actively find the target angles for dorsiflexion and plantar flexion separately, starting from the 0° point with their eyes closed. The margin of error between the reached angles and target angles will be recorded in degrees (°). Measurements will be repeated three times in the side-lying position for both ankles, and the average values will be recorded.
Isometric Muscle Strength | Through study completion, an average of 5 months
  The ankle dorsi flexor, plantar flexor, invertor and evertor isometric muscle strength will be measured using a digital dynamometer (Model-01165, Lafeyette Instrument®, USA) in the supine position, with the knee joint stabilised in extended position with the help of a belt. Three consecutive measurements will be recorded in kilogram and will be averaged. Thirty seconds rest intervals will be given between each measurement.
Static Balance | Through study completion, an average of 5 months
  The "Standing Stork Balance Test (SSBT)" will be used to assess static balance. The participant stands barefoot with their hands on their hips. They lift one leg and place the sole of the lifted foot against the inside of the opposite knee. The timer starts as soon as the participant is in position and stops when: The participant's heel touches the ground. The lifted foot moves away from the knee. The participant loses balance or moves their hands from their hips. Each participant will be performed the test three times and the average time for each leg was recorded as seconds for each sides.
Reaction Time | Through study completion, an average of 5 months
  Foot reaction time will be measured using the MoART (Multi-Operational Apparatus for Reaction Time) Lafayette Reaction Measuring device (Lafayette Instrument Company, Model no. 35601, USA), which is generally used for hand reaction assessments. In this study, the device will be modified for ankle reaction time measurements. For plantar flexor reaction time, the response mode will be set to "press," and for dorsiflexor reaction time, it will be set to "release." Three measurements will be taken for each test on both sides, and the average will be recorded in milliseconds (msec). All measurements will be performed in a quiet environment with participants seated on a back-supported chair.
Postural Stability | Through study completion, an average of 5 months
  The PROKIN-PK200W* (Tecnobody, Italy) device will be used to evaluate postural stability. Four different half-spherical heads can be placed under the mobile platform: easy/shallow, medium, hard/deep or rectangular. In the current study, two measurements will be taken in 30 seconds in bipedal stance with the hands on the waist using the easy head of the device and the average values will be recorded. A total of five different data will be obtained from the participants: total oscillation amount (circumference value), percentage value of the area gap showing the percentage of the area drawn according to the reference circle, oscillation speed, average oscillations in the antero-posterior (AP) and medio-lateral (ML) directions.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Miçooğulları, PhD, Principal Investigator — Cyprus International University
Locations (1):
- Cyprus International University, Mersin, Haspolat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Can be shared upon request.
Supporting Information: Study Protocol

REFERENCES:
- [Result] Park H, Kim KJ, Komatsu T, Park SK, Mutoh Y. Effect of combined exercise training on bone, body balance, and gait ability: a randomized controlled study in community-dwelling elderly women. J Bone Miner Metab. 2008;26(3):254-9. doi: 10.1007/s00774-007-0819-z. Epub 2008 May 11. PMID 18470666
- [Result] Sherrington C, Lord SR, Finch CF. Physical activity interventions to prevent falls among older people: update of the evidence. J Sci Med Sport. 2004 Apr;7(1 Suppl):43-51. doi: 10.1016/s1440-2440(04)80277-9. PMID 15214601
- [Result] Loureiro V, Gomes M, Loureiro N, Aibar-Almazan A, Hita-Contreras F. Multifactorial Programs for Healthy Older Adults to Reduce Falls and Improve Physical Performance: Systematic Review. Int J Environ Res Public Health. 2021 Oct 15;18(20):10842. doi: 10.3390/ijerph182010842. PMID 34682586
- [Result] Gillespie LD, Robertson MC, Gillespie WJ, Sherrington C, Gates S, Clemson LM, Lamb SE. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007146. doi: 10.1002/14651858.CD007146.pub3. PMID 22972103
- [Result] Toledo DR, Barela JA. Sensory and motor differences between young and older adults: somatosensory contribution to postural control. Rev Bras Fisioter. 2010 May-Jun;14(3):267-75. English, Portuguese. PMID 20730372
- [Result] He H, Luo C, Chang X, Shan Y, Cao W, Gong J, Klugah-Brown B, Bobes MA, Biswal B, Yao D. The Functional Integration in the Sensory-Motor System Predicts Aging in Healthy Older Adults. Front Aging Neurosci. 2017 Jan 5;8:306. doi: 10.3389/fnagi.2016.00306. eCollection 2016. PMID 28111548